CLINICAL TRIAL: NCT02754271
Title: Fit for Dialysis: Research-based Film as a Knowledge Translation Strategy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Toronto Rehabilitation Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Pia Kontos, Senior Scientist, Toronto Rehabilitation Institute
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 14-7507-DE
Record Dates: First submitted 2016-04-21; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: End-Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): A research-based film (Fit for Dialysis) and a 16-week exercise program involving activities during dialysis, at home, and in the community.
  Interventions: Other: Fit for Dialysis
- Control (No Intervention): The 16-week exercise program involving activities during dialysis, at home, and in the community.

INTERVENTIONS:
Other: Fit for Dialysis — A 15-minute research-based film that explores the barriers and facilitators regarding exercise participation by older hemodialysis patients and support by nephrology staff and family caregivers, and a 16-week exercise program involving activities during dialysis, at home, and in the community.
  Arms: Intervention

SUMMARY:
Exercise training for older hemodialysis patients can greatly improve many of the negative effects and poor health outcomes associated with end-stage kidney disease. Exercise has yet to be incorporated effectively and systematically into routine care. Exercise programs remain rare. When such programs are implemented, their participation rates vary, and they neglect home and community-based activities, as well as the involvement of family caregivers to support and reinforce exercise. This study is intended to address these limitations by introducing a highly accessible and compelling educational film, Fit for Dialysis, designed to introduce, motivate, and sustain exercise for wellness amongst older hemodialysis patients, and exercise counseling and support by family caregivers, nephrologists, and nurses. The objective of this clinical trial is to determine whether and in what ways Fit for Dialysis improves outcomes and influences knowledge/attitudes regarding the importance of exercise-based principles of wellness in the context of end-stage renal disease. Ultimately Fit for Dialysis could be used as a model for dialysis education that supports guideline recommendations that exercise be incorporated into the care and treatment of dialysis patients.

DETAILED DESCRIPTION:
The study introduces a highly accessible and compelling educational film designed to introduce, motivate, and sustain patient exercise for wellness amongst older hemodialysis patients, and exercise counseling and support by nephrology staff and family caregivers. Fit for Dialysis is a filmed drama that is based on focus group research with older hemodialysis patients, family caregivers, and health care practitioners that highlighted patients' desire to exercise as well as discouragement of patients to do so by overprotective families, and nurses' preferences for patient sedentariness during hemodialysis. Fit for Dialysis was tailored to the exigencies of out-patient hemodialysis settings by acknowledging and providing a roadmap to overcome the disciplinary silos and paternalism towards patients which inhibit exercise during hemodialysis, and highlighting some of the life circumstances that may influence patients' self-management of exercise behaviours at home and in the community.

In order to advance our understanding of the ways in which Fit for Dialysis influences participant outcomes, a prospective 2-site parallel intervention trial will be implemented that will compare the film + a 16-week exercise program in one hospital, with a 16-week exercise-only program in another hospital. Each hospital will have a 12-week follow-up. Qualitative and quantitative methods will be used including semi-structured interviews, and physical fitness and activity measures. These data will be used to explore the impact of Fit for Dialysis on: the knowledge/attitudes of patients, family caregivers, and staff regarding exercise-based principles of wellness; the education, motivation, or maintenance of patient exercise during dialysis, at home, and in the community; adherence to exercise prescription; and patient physical fitness and activity outcomes. The study will also explore factors related to family caregivers, nephrologists, nurses, and hospital administrators, and patients' home and community environments that may impact the successful uptake of the key messages of Fit for Dialysis.

In the intervention site (film+exercise hospital), 30 patients will view Fit for Dialysis and participate in the exercise program; at the exercise-only hospital, 30 patients will only exercise. A family caregiver of each participating patient will either view Fit for Dialysis and read an information letter on the benefits and contraindications of exercise (in the film+exercise hospital), or will only read the information letter (in the exercise-only hospital). In the film+exercise hospital, five nephrologists, 10 nurses and 3 administrators will also view the film. In both hospitals, 10 patients, 10 family caregivers, 10 nurses, 5 nephrologists, 3 administrators, and the physiotherapist assistants will be interviewed.

ELIGIBILITY:
Inclusion Criteria:

* Have conversational ability in English
* Have a medical diagnosis of hemodialysis-dependent end-stage renal disease
* Are a registered hemodialysis patient in the hospital for at least 3 months
* Receive ≥ 2 in-centre hemodialysis sessions per week
* Are ambulatory (with or without aids)
* Are deemed medically eligible by their nephrologist to participate in an exercise program that includes stretching, strengthening, and cardiovascular components
* Have a family caregiver who agrees to participate in the exercise program and keep a log of exercises on non-dialysis days

Exclusion Criteria:

* Currently participating in regular physical activity (structured exercise that includes a cardiovascular and/or strengthening component ≥ 3 times/week for ≥ 10 min/session

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-09 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Adherence measured by the percentage of time participants achieved at least 70% of prescribed targets of minutes and intensity of exercise per week. | 1-16 weeks
Change in functional exercise capacity measured by the 2-Minute Walk Test | 0, 8, 16, 28 weeks

SECONDARY OUTCOMES:
Change in number of steps using a pedometer | 0, 8, 16, 28 weeks
Change in basic mobility using the Timed Up and Go | 0, 8, 16, 28 weeks
Change in self-assessment of functional of capacities and peak metabolic equivalents using the Duke Activity Status Index | 0, 8, 16, 28 weeks
Change in upper extremity strength as a predictor of mortality and deteriorating health using the Grip Strength Test | 0, 8, 16, 28 weeks
Change in the frequency of mild, moderate, and strenuous bouts of exercise using the Godin Leisure-Time Exercise Questionnaire | 1-16, 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pia Kontos, PhD, Principal Investigator — University Health Network, Toronto
Locations (2):
- Canada (2):
  - Humber River Hospital - Wilson Site, Toronto, Ontario
  - St. Joseph's Health Centre - Satellite Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kontos P, Grigorovich A, Colobong R, Miller KL, Nesrallah GE, Binns MA, Alibhai SMH, Parsons T, Jassal SV, Thomas A, Naglie G. Fit for Dialysis: a qualitative exploration of the impact of a research-based film for the promotion of exercise in hemodialysis. BMC Nephrol. 2018 Aug 6;19(1):195. doi: 10.1186/s12882-018-0984-4. PMID 30081845
- [Derived] Kontos P, Alibhai SM, Miller KL, Brooks D, Colobong R, Parsons T, Jassal SV, Thomas A, Binns M, Naglie G. A prospective 2-site parallel intervention trial of a research-based film to increase exercise amongst older hemodialysis patients. BMC Nephrol. 2017 Jan 26;18(1):37. doi: 10.1186/s12882-017-0454-4. PMID 28122510